CLINICAL TRIAL: NCT03005171
Title: Perioperative Epidural Versus Intravenous Local Anesthetic Infusion in Open Upper Abdominal Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Mohamed Moatasem, Assistant Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00008718/1438
Record Dates: First submitted 2016-12-25; First posted 2016-12-29 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidural (Active Comparator): Epidural catheters will be placed in the 9th or 10th thoracic intervertebral space prior to induction of anesthesia.Through the thoracic epidural catheter 0.125% bupivacaine at a rate of 5 mL/h will be infused.
  The infusion continues for 24h
  Interventions: Drug: Bupivacaine
- Lidocaine (Active Comparator): Intravenous lidocaine infusion will typically start in the operating room prior to induction of anesthesia at a rate of 2 to 3 mg/min. Postoperatively, the rate will be decreased to 0.5 to 1 mg/min.
  The infusion continues for 24h
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Bupivacaine — Thoracic epidural bupivacaine infusion
  Other Names: Marcaine
  Arms: Epidural
Drug: Lidocaine — Intravenous lidocaine infusion
  Other Names: Xylocaine; Lidocaine Hydrochloride
  Arms: Lidocaine

SUMMARY:
The study evaluates the efficacy of intravenous lidocaine as an analgesic modality in patients undergoing open upper abdominal surgery; when compared with thoracic epidural analgesia. Half of participants will receive intravenous lidocaine infusion, while the other half will receive thoracic epidural bupivacaine infusion.

DETAILED DESCRIPTION:
Postoperative pain is one of the commonest problems encountered by anaesthesiologists, especially after open abdominal surgeries, in which post-operative pain would cause a restrictive respiratory dysfunction, which is associated with poor postoperative outcomes. Despite the fact that epidural blocks provide superior analgesia; it is not often an ideal option as it frequently causes hypotension that may require excessive intravenous fluid administration, which is particularly deleterious after bowel surgery. Other complications include epidural hematoma and higher failure rate. Furthermore epidural analgesia may be contraindicated in some patients e.g. patients on certain anti-platelet therapy and patients refusing the technique.

Other modalities to control postoperative pain are used e.g. intravenous analgesics and continuous wound infiltration, but none of which was proven to be as effective as epidural block.

Whether perioperative lidocaine infusion is as effective as epidural block in reducing post-operative pain, is this study's concern.

Some researches studied the efficacy of lidocaine infusion in controlling neuropathic as well as acute postoperative pain with encouraging results. Lidocaine infusion was found to reduce postoperative pain, opioid consumption and the length of hospital stay. Although risks of neurological and cardiac toxicity exist, these were not substantiated in the trials.

Lidocaine has been described to have both analgesic, and anti-hyperalgesic effects6, as well as anti-inflammatory properties. It also accelerates the return of post-operative gastrointestinal function, which is of particular importance after major abdominal surgery. Opposite to opioids, which increase the incidence of nausea and vomiting, lidocaine decreases their incidence.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open upper abdominal surgery

Exclusion Criteria:

* Bleeding diathesis
* History of allergy to local anesthetics
* Pregnancy/ lactation
* Cardiovascular disease
* Respiratory disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01; Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Verbal Numeric Rating Score | 2-24 hours
  Verbal Numeric Rating Score is an 11-point scoring system used to assesses the postoperative pain level of the participants

SECONDARY OUTCOMES:
B- endorphin level | Baseline-24 hours
  A measure for postoperative pain response compared to the baseline values
FVC | Baseline-24 hours
  Forced Vital Capacity
FEV1 | Baseline-24 hours
  Forced Expiratory Volume

CONTACTS AND LOCATIONS:
Overall Officials: Assiut University, Study Director — Assiut University, Egypt

IPD SHARING:
Plan to Share IPD: Undecided